CLINICAL TRIAL: NCT03595150
Title: Diclofenac for Prevention of Post-ERC Pancreatitis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Senior Consultant, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Post-ERCP-01
Record Dates: First submitted 2018-06-28; First posted 2018-07-23 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Common Bile Duct Diseases
Keywords: Endoscopic Retrograde Cholangiopancreatography; Pancreatitis; Diclofenac
MeSH Terms: conditions — Common Bile Duct Diseases; Pancreatitis | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: Open label randomised controlled trial of Diclofenac as prophylaxis versus no prophylaxis for prevention of post-ERCP pancreatitis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diclofenac (Active Comparator): 100 mg Diclofenac rectally prior to the ERCP
  Interventions: Drug: Diclofenac
- No prophylaxis (No Intervention): No prophylaxis

INTERVENTIONS:
Drug: Diclofenac — Diclofenac rectally given before the ERCP to prevent pancreatitis
  Arms: Diclofenac

SUMMARY:
The study aims at assessing the effectiveness of Diclofenac for prevention of post-ERCP pancreatitis. It will be undertaken embedded in the Swedish national register for Gallstone surgery and ERCP (GallRiks). Patients are randomised to Diclofenac prior to the ERCP or no prophylaxis. GallRiks is used to identify which patients fulfill the eligibility criteria and which patients develop pancreatitis after the ERCP.

DETAILED DESCRIPTION:
Endoscopic Retrograde Cholangiopancreatography (ERCP) is a procedure commonly performed for diagnosing changes in the bile ducts or managing outflow obstruction. Although ERCP may in most cases be performed safely, there is a risk of developing acute pancreatitis following the procedure. The risk has been estimated to 5-10%, with an increased risk in women, younger patients and in case the cannulation is difficult.

Phospholipase 2 is crucial in the pathogenesis of acute pancreatitis. As Diclofenac is a potent inhibitor of Phospholipase 2, it has been suggested that it may be used for prevention of post-ERCP pancreatitis. There is some evidence for the effectiveness of Diclofenac, but more studies are needed to confirm that it reduces the risk of post-ERCP pancreatitis.

In order to test whether Diclofenac reduces the risk for post-ERCP pancreatitis, a register-based randomized controlled study is planned. The study will be conducted embedded in the Swedish Register for Gallstone Surgery and ERCP (GallRiks). GallRiks includes data corresponding to the eligibility criteria as well as outcome measures. GallRiks will also be used to record which patients have been screened for inclusion.

Patients who meet the eligibility criteria are invited to the study. If they accept inclusion, they are randomized to 100 mg Diclofenac prior to the ERCP or np prophylaxis. No blinding is done.

The aim is to include 1000 patients. When 500 patients have been included, an interim analysis will be performed, comparing the incidence of pancreatitis and mortality in the two groups. A retrospective review of the patient records will be performed for those who develop pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ERCP

Exclusion Criteria:

* Decision to perform ERCP taken intraoperatively
* Intolerance/allergy against NSAID
* Patients taking NSAID daily
* Severe cardiac fail (ASA>4)
* Kidney failure (GFR<30 ml/min)
* Coagulation disorder
* History of peptic ulcer bleeding
* History of abdominoperineal resection
* Pregnancy
* Patients who do not understand Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis | Within 30 days post-ERCP
  Acute pancreatitis recorded in GallRiks by responsible endoscopist or surgeon. According to GallRiks criteria pancreatitis includes elevated amylase and abdominal pain of an intensity that hospital stay is warranted.

SECONDARY OUTCOMES:
Adverse drug reactions | Within 30 days post-ERCP
  Kidney failure, gastroduodenal ulcer or gastrointestinal bleeding
Mortality | Within 30 days post-ERCP
  Death within 30 days after ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, Ass Prof, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Undecided